CLINICAL TRIAL: NCT05624775
Title: Nourishing the Community Through Culinary Medicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Natalia Heredia, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-21-0555
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Culinary Medicine (Experimental)
  Interventions: Behavioral: Virtual Culinary Medicine

INTERVENTIONS:
Behavioral: Virtual Culinary Medicine — The virtual curriculum will include five 90-minute sessions (to be held weekly or bi-weekly). Participants will cook and engage virtually (with video and sound on) from their home kitchens via the digital platform. Participants will also be expected to shop for groceries ahead of the sessions to participate in the program. A gift card will be provided for groceries ($20 per class = $100 total).Asynchronous virtual educational content (cooking skills videos, animated nutrition education videos, and additional recipes) will be provided to engage and retain participants beyond initial sessions. Recipes will provide enough food for a family of four. clinic patients

SUMMARY:
The purpose of this study is to adapt existing Nourish Program curriculum for synchronous virtual delivery,to implement adapted virtual Culinary Medicine (CM)curriculum among target population, to assess if program participation improves participant dietary behaviors, nutrition knowledge, and cooking skills and behaviors above standard of care, to assess if program participation improves patient levels of HbA1c, Body Mass Index, Blood Pressure, HDL, LDL and Triglycerides above standard of care and to determine the feasibility and reproducibility of virtual synchronous CM classes in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes and glycosylated hemoglobin (HbA1c) >7.0
* receiving care at Sanitas Medical Center clinics in August 2021 - August 2023
* English speaking or Spanish speaking.

Exclusion Criteria:

* Patients without the technological support needed to participate in the program (e.g., reliable internet and device - cell phone, tablet or laptop);
* Patients with terminal or late-stage conditions (e.g., advanced stage chronic kidney disease);
* Patients with uncontrolled mental disorder that interferes with participation in active programming;
* Patients with physical impairment that interferes with participation in active programming

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Healthy Food Servings by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 3 items that are scored from 1 [None] to 6 [4 servings or more] for a maximum score of 18, a higher number indicating a better outcome.
Change in Typical food consumption behaviors by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 7 items that are scored from 1 [Not at all] to 5 [More than once a day] for a maximum score of 35, a higher number indicating better outcome.
Change in Perceived Barriers to Healthy Eating by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 9 items that are scored from 1 [Strongly Disagree] to 5 [Strongly Agree] for a maximum score of 45, a higher number indicating more perceived barriers.
Change in Shopping, cooking, and eating behaviors by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 9 items that are scored from 1 [Never] to 5 [Always], for a maximum score of 45, with a higher number indicating more ideal shopping, cooking and eating behaviors that align with program goals.
Change in Diabetes Management by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 18 items. The first 16 items that are scored from 1 [Does not apply to me] to 4 [Applies to me very much] and the remaining 2 items are dichotomous scored [Yes=1] to [No=0], for a maximum score of 68, with a higher number indicates a better diabetes self-management.
Change in cooking self-efficacy by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 10 items that are scored from 1 [Not sure at all] to 5 [Extremely sure], for a maximum of 50, with a higher number indicating more self-efficacy. Five items ask about self-efficacy before the program, and five ask about self-efficacy after the program.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)
Change in Body Mass Index | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)
Change in systolic Blood Pressure | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)
Change in diastolic Blood Pressure | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)
Change in High-density lipoprotein (HDL) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)
Change in low-density lipoprotein (LDL) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)
Change in Triglyceride | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion), and post 6-months completion of NCCM (within 90 days of 6-months completion of NCCM)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia I Heredia, PhD., MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No